CLINICAL TRIAL: NCT04030442
Title: Human Laboratory Model to Screen Drugs With Opioid Analgesic-sparing Effects: Cannabidiol/Morphine Combinations
Brief Title: Cannabidiol, Morphine, Pain
Acronym: CMP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Leslie Lundahl, Associate Professor, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CMP
Record Dates: First submitted 2019-06-17; First posted 2019-07-24 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: CBD; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smoked cannabidiol 0% (Placebo Comparator)
  Interventions: Drug: Immediate-release Oral Morphine Sulfate Tablets; Other: Thermal and Pressure Nociceptive Sensitivity
- Smoked cannabidiol 9.7% (Active Comparator)
  Interventions: Drug: Immediate-release Oral Morphine Sulfate Tablets; Other: Thermal and Pressure Nociceptive Sensitivity

INTERVENTIONS:
Drug: Immediate-release Oral Morphine Sulfate Tablets — 0 mg Immediate release oral morphine; 15 mg Immediate release oral morphine; 30 mg Immediate release oral morphine; Randomized between sessions
Other: Thermal and Pressure Nociceptive Sensitivity — Primary outcome measures of pain threshold and tolerance.

SUMMARY:
The purpose of the proposed study is to investigate the interaction of cannabidiol (CBD) and morphine effects on pain sensitivity. Cannabidiol is a cannabinoid (similar to cannabis, or marijuana) present in marijuana that alters some of the effects of marijuana.

DETAILED DESCRIPTION:
Eligible participants will be asked to participate in a total of three experimental sessions with each session day separated by at least one week. Each session day will last approximately 6-7 hours.

In the morning of each of the three study sessions, participants will be asked to complete baseline assessments which include self-report questionnaires (answering questions about how they feel), vital sign measurements (blood pressure, heart rate, oxygen saturation, temperature, and pupillometry) will be taken using a non-invasive (external) vitals monitor, and lastly thermal (heat and cold) and mechanical sensitivity testing will be done.

Participants will be asked to take an oral morphine capsule.

Participants will participate in 2 smoking sessions where they will be asked to smoke cigarettes or a vaporizer balloon containing either cannabidiol or a placebo (a blank).

Participants will be asked to complete the same battery assessments mentioned above, which include self-report questionnaires (answering questions about how they feel); vital sign measurements (blood pressure, heart rate, oxygen saturation, temperature, and pupillometry) will be taken using a non-invasive (external) vitals monitor; and lastly thermal (heat and cold) and mechanical stimulation will be administered to test pain sensitivity.

Participants will be asked to complete subjective questionnaires and have vital signs (blood pressure, heart rate, oxygen saturation, temperature, and pupillometry) measured multiple times throughout the visit; these measurements will be monitored for reasons such as safety.

After completing the second round of smoking and battery assessments, participants will be provided with lunch and can relax, watch television, listen to music, or read.

Once vital signs and questionnaire ratings have returned to baseline levels; participants can leave the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Participants must report having smoked a cigarette (nicotine or marijuana) AND having taken an opioid on 3 or more occasions in their lifetime.
* Participants must be in good health to participate; those with certain contraindications will be excluded.
* All participants will undergo psychiatric evaluation and will be asked to report their substance use history by interview and structured questionnaire methods.
* Participants will undergo medical evaluations using medical history, physical exam, standard lab tests (complete blood chemistry, urinalysis, urine pregnancy test for females), and 12-lead ECG.

Exclusion Criteria:

* Serious psychiatric illness (e.g. psychotic or bipolar disorder, recent suicide attempts; severe depression)
* Substance Use Disorders other than Nicotine Use Disorder and Mild Cannabis Use Disorder
* Neurological diseases; cardiovascular problems (e.g. systolic BP >140 or <95 mmHg, diastolic BP >90 mmHg, abnormal ECG); pulmonary diseases; systemic diseases (e.g. liver, renal, inflammatory)
* Cognitive impairment (<80 IQ)
* Past-month medications that increase study risk
* Women who are pregnant (urine HCG), lactating (self-report), or if heterosexually active and not using (self-report) medically approved birth control (oral or depot contraception, IUD, condom/foam, sterilization, tubal ligation)
* Individuals unable to give informed consent will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-01-26 (Estimated); Study Completion 2025-01-26 (Estimated)

PRIMARY OUTCOMES:
CHANGE: PAIN THRESHOLD AND TOLERANCE Pain responses to a range of heat, cold and mechanical pressure stimuli | Pain responses measured at the start of the visit, baseline; 25 minutes post CBD 0% drug; 25 minutes post CBD 9.7% drug
  Change in pain threshold and tolerance is being assessed post each CBD drug use (0%and 9.7%) using Q-Sense Conditioned Pain Modulation™. A randomized series of 7 heat stimuli and 7 cold stimuli will be delivered via a thermode attached to the lower nondominant arm. A series of 7 pressure stimuli will be delivered with a pressure algometer to the opposite arm.

SECONDARY OUTCOMES:
SAFETY: Systolic blood pressure (physiological effects) | Systolic blood pressure measured at baseline; 30 and 45 minutes post-morphine; 15 minutes post CBD 0% drug; 15, 65, and 90 minutes post 9.7% CBD drug (final drug).
  Safety is being assessed.
SAFETY: Diastolic blood pressure (physiological effects) | Diastolic blood pressure measured at baseline; 30 and 45 minutes post-morphine; 15 minutes post CBD 0% drug; 15, 65, and 90 minutes post 9.7% CBD drug (final drug).
  Safety is being assessed.
SAFETY: Heart rate | Heart Rate measured at baseline; 30 and 45 minutes post-morphine; 15 minutes post CBD 0% drug; 15, 65, and 90 minutes post 9.7% CBD drug (final drug).
  Safety is being assessed.
SAFETY: Temperature | Temperature measured at baseline; 30 and 45 minutes post-morphine; 15 minutes post CBD 0% drug; 15, 65, and 90 minutes post 9.7% CBD drug (final drug).
  Safety is being assessed.
SAFETY: Oxygen saturation | Oxygen Saturation measured at baseline; 30 and 45 minutes post-morphine; 15 minutes post CBD 0% drug; 15, 65, and 90 minutes post 9.7% CBD drug (final drug).
  Safety is being assessed.
SAFETY: Pupillometry Measurement - Diameter of your eye | Pupillometry measured at baseline; 30 and 45 minutes post-morphine; 15 minutes post CBD 0% drug; 15, 65, and 90 minutes post 9.7% CBD drug (final drug).
  Safety is being assessed.
SAFETY & INDICES OF ABUSE LIABILITY: Drug Effect | Drug Liking measured at baseline; 30 and 45 minutes post-morphine; 15 minutes post CBD 0% drug; 15, 65, and 90 minutes post 9.7% CBD drug (final drug).
  Indices of abuse liability is being assessed. Visual Analog Scales (0="not at all" and 100= "extremely"): "good drug effect," "bad drug effect," "strength of drug effect," liking," "sedated," "high" and "desire to take again."
SAFETY & INDICES OF ABUSE LIABILITY: Drug Symptoms | Drug Symptoms measured at baseline; 30 and 45 minutes post-morphine; 15 minutes post CBD 0% drug; 15, 65, and 90 minutes post 9.7% CBD drug (final drug).
  Drug Symptoms are being assessed, (0="not at all", 1= "a little", 2="moderately", 3="quite a bit" 4= "extremely").
SAFETY & INDICES OF ABUSE LIABILITY: Mood and Feeling | Measured at baseline; 30 and 45 minutes post-morphine; 15 minutes post CBD 0% drug; 15, 65, and 90 minutes post 9.7% CBD drug (final drug).
  Mood and Feeling is being assessed. Visual Analog Scales (0="not at all" and 100= "extremely"): "Anxious", "Sedated", "Hungry", "Stimulated", "Friendly", "High", "Alert", "Happy", "Tired", "Talkative", "Self-Confident", "Down", "Social", "Upset", "Confused", "Good Drug Effect", "Bad Drug Effect", "Dizzy", "Sleep", "Energetic", "Jittery", "Content", "Unmotivated", "Restless", "Forgetful", "Mellow", "Clumsy", "Numbness or tingling in my extremities", "I'm having difficulty concentrating", "I am sweating", "My heart is pounding or beating faster than usual", "Noises or sounds seem louder than usual", "My limbs feel heavier than usual".
SAFETY & INDICES OF ABUSE LIABILITY: Feelings about self | Measured at baseline; 30 and 45 minutes post-morphine; 15 minutes post CBD 0% drug; 15, 65, and 90 minutes post 9.7% CBD drug (final drug).
  One's self-evaluation of feelings is being assessed.
SAFETY & INDICES OF ABUSE LIABILITY: Brief Pain Inventory | Measured at baseline only.
  One's self-evaluation of pain is being assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Lundahl, PhD, Principal Investigator — Wayne State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States